CLINICAL TRIAL: NCT06639061
Title: Characterization and Modulation of Traumatic Memories in PTSD Patients Using Transcranial Magnetic Stimulation (TMS)
Brief Title: Neuromodulation of the Hippocampus to Reduce Intrusive Re-Experiencing in PTSD: A Randomized Controlled Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Yair Bar-Haim, Professor, Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0004373-5; 101141436 - TraumaNeuroInsight (Other Grant/Funding Number: European Research Council (ERC))
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: PTSD - Post Traumatic Stress Disorder; Intrusive Memories of Traumatic Event(s)
Keywords: PTSD; TMS; MRI
MeSH Terms: conditions — Combat Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Trauma memory reactivation + targeted hippocampal TMS (Active Comparator): Brain stimulation using repetitive transcranial magnetic stimulation (rTMS) will be given after a deliberate memory re-activation, using repetitive pulses at 1Hz frequency for 15 minutes, once a week over 5 weeks. The scalp stimulation area will be determined based on a resting state fMRI scan identifying a cortical area that is most strongly functionally connected to the left hippocampal target of each patient.
  Interventions: Device: Hippocampal stimulation using repetitive transcranial magnetic stimulation (rTMS)
- Trauma memory reactivation + targeted sham TMS (Sham Comparator): Brain stimulation using repetitive transcranial magnetic stimulation (rTMS) will be given after a deliberate memory re-activation, using repetitive pulses at 1Hz frequency for 15 minutes, once a week over 5 weeks. The scalp stimulation area will be determined based on a resting state fMRI scan identifying a cortical area that has near zero functional connectivity with the left hippocampal target of each patient.
  Interventions: Device: Sham stimulation using repetitive transcranial magnetic stimulation (rTMS)

INTERVENTIONS:
Device: Hippocampal stimulation using repetitive transcranial magnetic stimulation (rTMS) — We will use fMRI resting state data to personalize a TMS inhibitory stimulation to a cortical location that is the most strongly connected to a deeper left hippocampal target.
  5 once a week sessions of rTMS will be delivered at 1-Hz stimulation frequency for 15 minutes following trauma memory reactivation.
  Other Names: TMS; MRI
  Arms: Trauma memory reactivation + targeted hippocampal TMS
Device: Sham stimulation using repetitive transcranial magnetic stimulation (rTMS) — We will use fMRI resting state data to personalize a TMS sham stimulation to a cortical location with near zero connectivity to a deeper left hippocampal target. 5 once a week sessions of rTMS will be delivered at 1-Hz stimulation frequency for 15 minutes following trauma memory reactivation.
  Other Names: TMS; MRI
  Arms: Trauma memory reactivation + targeted sham TMS

SUMMARY:
The goal of this clinical trial is to learn if non-invasive neurostimulation of memory-related brain areas works to treat intrusive memory symptoms in adults patients with posttraumatic stress disorder (PTSD). It will also learn about the effect of this neuromodulation procedure on reorganization of memory-related brain networks. The main questions it aims to answer are:

Does neuromodulation lower the number of times and the emotional severity participants intrusive memories? Does neuromodulation reduces the overall severity of PTSD? Researchers will compare neuromodulation targeting the hippocampus (a memory-related brain structure) to a control stimulation in an area not related to memory processes to see if hippocampus neuromodulation works to treat intrusive trauma memories and PTSD.

Participants will:

1. Undergo magnetic resonance imaging (MRI) scans before and after neuromodulation to: a) determine a personalized neuromodulation target; and b) to measure changes in brain function from before to after treatment.
2. Receive hippocampus neuromodulation or a control neuromodulation once a week for 5 weeks.

Keep a daily diary of their symptoms and the number of times they experience intrusive trauma memories.

DETAILED DESCRIPTION:
Intrusive trauma memories are a hallmark of posttraumatic stress disorder (PTSD), and the least treatment responsive. Thus, revealing neurocognitive mechanisms associated with intrusive trauma memories has been indexed a priority. Prior work shows that targeting hippocampal circuitry modulates functional connectivity among distributed cortical-hippocampal network regions and alters memory performance in healthy participants. In the current clinical trial we test hypotheses on the clinical effects of such stimulation in a two-arms randomized controlled trial: Trauma memory reactivation + targeted hippocampal transcranial magnetic stimulation TMS (R-H-TMS) and Trauma memory reactivation + Control TMS (over the SMA; R-C-TMS). We will test a) Hippocampus seed-based connectivity patterns - revealing the impact of the targeted stimulation on extended memory brain networks; and b) frequency and severity of intrusive memory symptoms. The R-H-TMS vs. R-C-TMS contrast will speak to specificity of the noted effects to hippocampal stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Aged of 20-65 years.
* Meet a diagnosis of PTSD according to DSM-5 as tested by a structured clinical interview (Clinician-Administered PTSD Scale for DSM-5 - CAPS-5).
* CAPS-5 total score greater or equal to 33.
* Endorsement of intrusive symptoms (flashbacks, nightmares, or intrusive memories) with a frequency of at least 3 times a week.
* Meeting the accepted criteria for inclusion in an MRI examination.

Exclusion Criteria:

* Meeting a diagnosis of Complex PTSD or personality disorder.
* Psychotic disorder, bipolar disorder, or a developmental neuropsychological disorder (autism, mental retardation).
* Use of psychiatric medications (except for the medications listed in section 4.a of the study protocol if the medication dosage is stable in the last three months and does not change during the study.
* Exclusion rules in TMS research (see guidelines).
* Use of the following drugs: imipramine, amitriptyline, doxepin, nortriptyline, maprotiline, chlorpromazine, clozapine, foscarnet, ganciclovir, ritonavir, amphetamines, cocaine, (MDMA, ecstasy), phencyclidine (PCP, angel's dust), ketamine, gamma- hydroxybutyrate (GHB), alcohol, theophylline
* Epilepsy or use of anti-epileptic drugs.
* Traumatic head injuries or head surgery.
* Implanted metallic body (except fillings/amalgam bites/orthodontic fixations approved for MRI), electrodes or a pacemaker.
* Migraines
* Pregnant women
* Hearing problems
* Drinking alcohol 24 hours before the TMS session
* Repeated episodes of fainting with loss of consciousness and/or an event of fainting with loss of consciousness in the past year.
* The accepted exclusion criteria for an MRI examination

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total score | Baseline, 6 weeks, 3-months
  The CAPS-5 is a 30-item structured interview that can be used to make current (past month or week) diagnosis of PTSD & make lifetime diagnosis of PTSD.

SECONDARY OUTCOMES:
PTSD Checklist for DSM-5 (PCL-5) | Baseline, 6 weeks, 3-months
  The PCL-5 is a 20-item self-reported measured based on the DSM-5 PTSD symptoms and assessing PTSD symptoms endorsement and severity.
Intrusive trauma memories diary | Through study completion, an average of 8 weeks
  The amount, frequency and emotional effect of intrusive traumatic memories, measured by a daily self-report digital diary.
Patient Health Questionnaire - 9 (PHQ-9) | Baseline, 6 weeks, 3-months
  Measures severity of depression symptoms as listed in the DSM-5

OTHER OUTCOMES:
credibility/expectancy questionnaire (CEQ) | Baseline
  Measures treatment expectancies and credibility
fMRI Neuroimaging | Baseline, 6 weeks
  Functional connectivity, indicating the level of synchronous activity of certain brain regions during rest (temporal correlation is usually expressed as a Pearson's r). Derived from the fMRI scans, and compared between the two groups as a function of time.

CONTACTS AND LOCATIONS:
Overall Officials: Yair Bar-Haim, PhD, Principal Investigator — Tel Aviv University
Locations (1):
- Tel Aviv University, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Yes
De-identified data from the study will be shared in accordance with local laws related to patient data sharing.
Supporting Information: Study Protocol, SAP
Time Frame: Uploaded by October 2026 (before data analyses starts), will stay on.
Access Criteria: Deidentified clinical outcome data will be deposited in an open access repository in compliance with local patient information sharing laws. Reference to the repository will be embedded in the published report for unrestricted access.
  De-identified MRI data matrices will be shared upon request and in compliance with local patient information sharing laws.